CLINICAL TRIAL: NCT00330707
Title: A Multi-centre Randomised Controlled Double-blinded Trial of BCG and Interferon Alpha in High Risk Superficial Bladder Cancer
Brief Title: Combined Use of BCG and Interferon Alpha in Bladder Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NMRC/0085/1995
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Carcinoma of Urinary Bladder, Superficial
Keywords: bladder cancer; BCG; interferon alpha
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — BCG Vaccine; Interferon-alpha

INTERVENTIONS:
Drug: Bacillus Calmette Guerin and interferon alpha

SUMMARY:
To compare the toxicity and efficacy of the combination of BCG and interferon alpha to standard dose and low dose BCG alone in high risk superficial bladder cancer

DETAILED DESCRIPTION:
140 eligible patients with high risk superifical bladder cancer would be randomised to receive standard dose BCG, low dose BCG or the combination of low dose BCG and interferon alpha in a schedule of "6+3" weekly intravesical instillations. Patients would be closely monitored with cystoscopy and urine cytology and intravenous urograms when indicated. Pre-and post-instillation urine samples would be collected for cytokine analysis.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients must have completely resected, histologically?proven urothelial carcinoma of the urinary bladder, stage Ta or Tl 1 ? 16 weeks prior to registration, and/or carcinoma-in-situ on bladder biopsy. Central pathology review was mandatory. (2) Patients with Stage Ta urothelial carcinoma must be judged to be at increased risk of tumor recurrence by virtue of any one of the following: (a) Tumor recurrence during the 56 weeks prior to registration, (b) Two or more initial tumors within 28 weeks, (c) Grade III urothelial carcinoma during the 16 weeks prior to registration, (d) Dysplasia or carcinoma-in-situ on random biopsy or (e) Positive urinary cytology post tumor resection. "Suspicious" or "suggestive" cytology is insufficient for this criterion. (3) Patients who have received prior intravesical therapy other than BCG were eligible provided they had not undergone a course of any other intravesical agent within two months prior to entry. (4) There was no age restriction; however, all patients registered had to be willing to be available for 5?year follow up and to have a life expectancy of at least two years. (5) Patients had a Karnofsky score >50. (6) Women of child?bearing age were using effective contraceptive methods. (7) Patients agreed not to take vitamin supplements (except for those prescribed in the study) for the duration of the trial. (8) Pretreatment laboratory tests and radiological examinations must have been obtained during the 16 weeks prior to patient registration. (9) All patients had to be informed of the investigational nature of this study, and had to sign a written informed consent in accordance with institutional guidelines.

Exclusion Criteria:

* (1) Patients with medical illness or mental status, which would preclude cooperation with the study. (2) Patients who were immunodeficient, or had received immunosuppressive radiation therapy or chemotherapy. (3) Patients with urothelial carcinoma of stage T2 or higher. (4) Patients who had evidence of urothelial carcinoma of the upper urinary tract at the time of recruitment. (5) Patients who had received radiation therapy for bladder cancer within one year prior to registration. (6) Patients who had been previously treated with intravesical BCG. (7) Patients with active tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 1995-10; Study Completion 2005-06

PRIMARY OUTCOMES:
local toxicity
systemic toxicity
recurrence rate
progression rate
disease-specific mortality

CONTACTS AND LOCATIONS:
Overall Officials: Kesavan Esuvaranathan, FRCSEd MD, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Chiong E, Kesavan A, Mahendran R, Chan YH, Sng JH, Lim YK, Kamaraj R, Tan TM, Esuvaranathan K. NRAMP1 and hGPX1 gene polymorphism and response to bacillus Calmette-Guerin therapy for bladder cancer. Eur Urol. 2011 Mar;59(3):430-7. doi: 10.1016/j.eururo.2010.11.031. Epub 2010 Dec 1. PMID 21163569